CLINICAL TRIAL: NCT07366853
Title: Feasibility and Safety of Intraneural Sciatic Nerve Block Via Lateral Mid-femoral Approach: A Clinical Study
Brief Title: Feasibility and Safety of Sciatic Nerve Paraneural Sheath Block Using a Mid-Femoral Lateral Approach
Acronym: iSNB-LF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Yan Ren-2026-01
Record Dates: First submitted 2026-01-08; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Adverse Effect; Feasibility Study; Safety and Effectiveness
Keywords: Sciatic Nerve Block; Subparaneural Block; Lateral Mid-femoral Approach; Popliteal Approach; Ultrasound-guided; Feasibility; Safety

STUDY DESIGN:
Intervention Model Description: This is a prospective, parallel-group, randomized, controlled, double-blinded (participant and outcome assessor), exploratory feasibility trial. It compares ultrasound-guided subparaneural sciatic nerve block via a novel lateral mid-femoral approach (experimental) with the conventional popliteal approach (active control) in patients undergoing below-knee surgery. The primary aim is to assess the feasibility and safety of the new approach. Participants are randomized 1:1. Blinding is achieved through general anesthesia (participant) and use of an independent, blinded assessor for outcome evaluation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral Mid-femoral Approach Sciatic Nerve Block (Experimental): Ultrasound-guided sciatic nerve subparaneural sheath block via the lateral mid-femoral approach. Under combined ultrasound and nerve stimulator guidance, a single injection of 20 mL of 0.5% ropivacaine hydrochloride will be administered into the paraneural sheath at the mid-femoral level.
  Interventions: Procedure: Ultrasound-guided lateral mid-femoral sciatic nerve block
- Popliteal Approach Sciatic Nerve Block (Active Comparator): Ultrasound-guided sciatic nerve subparaneural sheath block via the conventional popliteal approach. Under combined ultrasound and nerve stimulator guidance, a single injection of 20 mL of 0.5% ropivacaine hydrochloride will be administered into the paraneural sheath at the popliteal fossa (prior to nerve bifurcation).
  Interventions: Procedure: Ultrasound-guided popliteal sciatic nerve block

INTERVENTIONS:
Procedure: Ultrasound-guided lateral mid-femoral sciatic nerve block — Ultrasound-guided sciatic nerve subparaneural sheath block via the lateral mid-femoral approach. Under combined ultrasound and nerve stimulator guidance, a single injection of 20 mL of 0.5% ropivacaine hydrochloride will be administered into the paraneural sheath at the mid-femoral level
  Arms: Lateral Mid-femoral Approach Sciatic Nerve Block
Procedure: Ultrasound-guided popliteal sciatic nerve block — Ultrasound-guided sciatic nerve subparaneural sheath block via the conventional popliteal approach. Under combined ultrasound and nerve stimulator guidance, a single injection of 20 mL of 0.5% ropivacaine hydrochloride will be administered into the paraneural sheath at the popliteal fossa (prior to nerve bifurcation).
  Arms: Popliteal Approach Sciatic Nerve Block

SUMMARY:
This study is designed as a randomized controlled trial aiming to evaluate the feasibility and safety of ultrasound-guided mid-femoral lateral approach sciatic nerve paraneural sheath block, in order to provide a new sciatic nerve block approach for clinical practice that offers greater patient comfort and higher precision, thereby facilitating its use for specific patient populations and less experienced operators.

DETAILED DESCRIPTION:
In clinical practice, the popliteal approach to sciatic nerve paraneural sheath block is the most commonly used. Studies have found that compared with extraneural injection, ultrasound-guided sciatic nerve paraneural sheath block via the popliteal approach has a faster onset and provides longer postoperative sensory and motor blockade. Paraneural sheath block aims to achieve efficient, rapid, and precise nerve blockade using a low volume of local anesthetic. However, the popliteal approach requires knee flexion for performance, necessitating the patient to be in a prone or lateral decubitus position. For patients unable to flex the knee or those with positioning difficulties due to conditions such as lower limb fractures, this method is less applicable. For the above reasons, the popliteal sciatic nerve block has certain limitations.

The mid-femoral lateral approach demonstrates unique advantages: First, the patient can maintain a supine position throughout the procedure, significantly enhancing comfort and compliance. Second, the sciatic nerve is relatively superficial at this level, offering good ultrasonographic visualization and being distant from major blood vessels and nerves. This makes it applicable even in obese patients with thick subcutaneous fat and suboptimal ultrasound images, theoretically enhancing procedural safety. Therefore, it is considered an effective solution for patients with positioning restrictions, such as those with lower limb fractures and severe pain, holding high potential for clinical promotion and research significance.

Although the anatomical feasibility of this approach has been preliminarily confirmed, its practical feasibility and safety require validation through clinical studies. In particular, whether a successful "paraneural sheath block" can be consistently achieved at the mid-femoral lateral level, similar to the classic popliteal approach, remains to be explored. While some literature suggests its theoretical feasibility, there is a lack of prospective, systematic clinical research evidence to support its practical application feasibility (e.g., block efficacy, procedural difficulty, success rate) and safety (e.g., complication rates, incidence of nerve injury).

This study is designed as a randomized controlled trial aiming to evaluate the feasibility and safety of ultrasound-guided mid-femoral lateral approach sciatic nerve paraneural sheath block. The goal is to provide a new sciatic nerve block option for clinical practice that offers greater patient comfort and more precise blockade, facilitating its use for specific patient populations and less experienced operators.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective unilateral surgery below the knee (e.g., internal fixation for ankle, metatarsal, or calcaneal fractures; hallux valgus correction; flatfoot reconstruction).
2. American Society of Anesthesiologists (ASA) physical status class I or II.
3. Aged 18 to 65 years.
4. Ability to understand the study procedure and provide written informed consent.

Exclusion Criteria:

1. Contraindications to peripheral nerve block:

   * Known allergy or history of toxicity to local anesthetics.
   * Pre-existing neuropathy in the operative limb.
   * Severe coagulopathy.
   * Infection at the intended needle puncture site.
   * Systemic infection.
2. Requirement for simultaneous surgery at a site other than the unilateral lower limb below the knee.
3. Previous surgery or significant scarring in the area of the planned needle insertion for the sciatic nerve block.
4. Body mass index (BMI) > 35 kg/m².
5. Patients receiving chronic pain therapy or with a history of opioid abuse.
6. Inability to communicate or cooperate with the study assessments (e.g., due to cognitive impairment, language barrier, or psychiatric disorder).
7. Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complete sensory blockade in the sciatic nerve distribution at 30 minutes after block completion | At 30 minutes after completion of the local anesthetic injection.
  The proportion of patients achieving complete sensory blockade (Grade III: numbness, no sensation to pinprick) in the tibial and common peroneal nerve distributions at 30 minutes following the administration of the local anesthetic. Sensory blockade will be assessed using von Frey filaments and compared to the contralateral limb.

SECONDARY OUTCOMES:
Block Success Rate | At 30 minutes after block completion.
  Proportion of patients achieving both complete sensory blockade (Grade III) and complete motor blockade (Grade III) in the sciatic nerve distribution at 30 minutes after local anesthetic injection.
Sensory Block Onset Time | From the end of injection until complete sensory block is achieved (assessed every 30 seconds), up to 30 minutes.
  Time interval from the end of local anesthetic injection to the achievement of complete sensory blockade (Grade III).
Duration of Sensory Block | From block onset until first pain complaint, assessed up to 48 hours postoperatively.
  Time interval from the onset of complete sensory blockade to the first complaint of pain in the surgical area (NRS > 0).
Motor Block Onset Time | From the end of injection until complete motor block is achieved (assessed every 30 seconds), up to 30 minutes.
  Time interval from the end of local anesthetic injection to the achievement of complete motor blockade (Grade III: inability to move the ankle).
Duration of Motor Block | From block onset until full motor recovery, assessed up to 48 hours postoperatively.
  Time interval from the onset of complete motor blockade to the recovery of normal ankle flexion and extension.
Time to First Request for Rescue Analgesia | From end of surgery until first rescue request, assessed up to 24 hours postoperatively.
  Time interval from the end of surgery to the patient's first activation of the patient-controlled intravenous analgesia (PCIA) pump or request for supplemental analgesia.
Total Consumption of Rescue Analgesics within 24 Hours | Within 24 hours after surgery.
  Total dose of rescue analgesics (e.g., parecoxib, ketorolac, morphine) administered within the first 24 postoperative hours.
Postoperative Pain Intensity (NRS Scores) | At 4, 8, and 24 hours after surgery.
  Pain intensity assessed using the Numerical Rating Scale (NRS, 0-10) at rest and during movement at 4, 8, and 24 hours postoperatively.
Incidence of Rebound Pain | Within 48 hours after block resolution.
  Proportion of patients experiencing rebound pain, defined as an NRS score >7 within 48 hours after block resolution, not relieved by multiple PCIA boluses within 30 minutes.
Procedure-Related Times | During the block procedure.
  1. Ultrasound Scanning Time: Time from probe placement to clear identification of the target nerve.
  2. Total Needle Manipulation Time: Time from needle insertion to completion of drug injection.
Number of Needle Redirections | During the block procedure.
  Total number of times the nerve stimulation needle is adjusted or redirected to achieve the final position.
Incidence of Complications | From block procedure up to 1 week postoperatively.
  Proportion of patients experiencing block-related complications, including local anesthetic systemic toxicity, nerve injury (persistent neuropathy), hematoma, or infection.
Patient Satisfaction Score | At 24 hours postoperatively.
  Patient-reported satisfaction with the overall anesthesia and analgesia experience, assessed using a 5-point Likert scale (0=very dissatisfied, 5=very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No